CLINICAL TRIAL: NCT03584737
Title: Multi-Center Study of a Point-of-Care Immunoassay for the Detection of Bacterial Sinusitis
Brief Title: Point-of-Care Immunoassay for Detection of Bacterial Sinusitis
Status: Terminated | Type: Observational
Why Stopped: Lack of funding
Sponsor: ENTvantage Dx (Industry)
Collaborators: Beaufort (Unknown)
Responsible Party: Sponsor
Other Study IDs: 1001
Record Dates: First submitted 2018-06-19; First posted 2018-07-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Sinusitis Bacterial
Keywords: acute sinusitis; bacterial sinusitis; point-of-care; in vitro diagnostic device (IVD)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — nasal mucus in buffer solution
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Symptomatic for bacterial sinusitis: Samples from participants showing symptoms of bacterial sinusitis tested by rapid in vitro diagnostic test, bacterial culture, and PCR assay
  Interventions: Diagnostic Test: rapid in vitro diagnostic test; Diagnostic Test: bacterial culture; Diagnostic Test: PCR assay

INTERVENTIONS:
Diagnostic Test: rapid in vitro diagnostic test — IVD for qualitative detection of 3 bacterial pathogens (Haemophilus influenzae, Moraxella catarrhalis, and Streptococcus pneumoniae)
  Other Names: Sinu-Test®
Diagnostic Test: bacterial culture — Quantitative bacterial culture assay with isolate identification by MALDI-TOF.
Diagnostic Test: PCR assay — Semiquantitative real-time PCR assay

SUMMARY:
This study is conducted to evaluate the performance of a rapid, point-of-care in vitro diagnostic device (Sinu-Test®) for the qualitative detection of the three most common pathogens responsible for causing bacterial sinusitis.

DETAILED DESCRIPTION:
Mucous specimens will be collected from patients displaying symptoms of acute bacterial sinusitis enrolled by primary care and/or otolaryngology clinics in the United States. Health care professionals not having endoscopy certification will collect specimens using the Entvantage sample collection device. Health care professionals with nasal endoscopy certification or specialty training will collect comparator specimens using an endoscope. Untrained operators with a range of education and training (primary care physician, otolaryngologist, physician assistant, nurse practitioner, registered nurse or other healthcare professional), will perform the Sinu-Test® lateral flow assay in an outpatient setting. Mucous samples will be tested for the presence of 3 bacterial pathogens responsible for sinusitis using the Sinu-Test® in the clinic and by a composite comparator method comprised of standard quantitative bacterial culture with identification (matrix-assisted laser desorption/ionization-Time of Flight (MALDI-TOF) mass spectrometry instrument) and semiquantitative real-time polymerase chain reaction (real-time PCR) of the residual culture sample and the Sinu-Test® residual swab performed by a central laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Meets definition of acute sinusitis by Infectious Disease Society of America (2012)

Exclusion Criteria:

* Chronic sinusitis
* Cystic fibrosis
* Patients treated with antibiotics currently or within the previous 30 days.
* Subjects with a prior history of sinus surgery will be excluded due to the modification of sinonasal anatomy.
* Primary immunodeficiencies, as self-reported

  * Combined variable immunodeficiency
  * Immunodeficiency with reduced immunoglobulin G (IgG) and immunoglobulin A (IgA)-bearing cells
  * Kartagener Syndrome (ciliary dyskinesia)
  * Agammaglobulinemia
  * Sickle cell disease
* Acquired immunodeficiencies, as self-reported

  * Chemotherapy
  * Radiation therapy
  * Transplantation
  * Asplenia
  * HIV
  * Poorly controlled Diabetes mellitus
* Cognitive impairment resulting in the inability to provide informed consent.
* Special groups, such as children under the age of 18, and men and women who are in prison will not participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at least 18 years of age with symptoms of bacterial sinusitis from primary care clinics and otolaryngology clinics.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2021-11-12 (Actual); Primary Completion 2023-04-09 (Actual); Study Completion 2023-04-10 (Actual)

PRIMARY OUTCOMES:
Sensitivity (positive predictive agreement) and specificity (negative predictive agreement) of the diagnostic device | Cumulation of one-time subject sample results obtained in 20-30 minutes for point-of-care test and 3-5 days for lab results
  Assessment of the true positive and true negative rate of the point-of-care test device relative to the composite reference standard for each of the 3 bacterial microorganisms.

SECONDARY OUTCOMES:
Positive predictive value (PPV) and negative predictive value (NPV) | Cumulation of one-time subject sample results obtained in 20-30 minutes for point-of-care test and 3-5 days for lab results
  Positive predictive value is the probability that subjects with a positive point-of-care test truly have the bacteria present. Negative predictive value is the probability that subjects with a negative point-of-care test truly do not have the bacteria present.
Positive likelihood ratio (LR+) and negative likelihood ratio (LR-) | Cumulation of one-time subject sample results obtained in 20-30 minutes for point-of-care test and 3-5 days for lab results
  LR+ is equivalent to the probability of a true positive result divided by the probability of a false positive result. LR- is equivalent to the probability of a false negative result divided by the probability of a true negative result.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Busch, Study Director — Beaufort
Locations (7):
- United States (7):
  - Northern California Research, Sacramento, California
  - Hillcrest Medical Research, DeLand, Florida
  - ENT Allergy & Associates of South Florida, Port Saint Lucie, Florida
  - Tandem Clinical Research, Marrero, Louisiana
  - Northwell Health, New Hyde Park, New York
  - Optimed Research/Ohio Sinus Institute, Dublin, Ohio
  - Kelsey-Seybold Clinic, Houston, Texas

IPD SHARING:
Plan to Share IPD: No